CLINICAL TRIAL: NCT04791046
Title: Personalized Evidence-based Medicine Improves Outcomes of Antihypertensive Therapy in Patients With Comorbidities
Brief Title: Antihypertensive Therapy in Patients With Comorbidities
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Center of Personalized Medicine, Pirogova (Other)
Collaborators: Center for New Medical Technologies, Novosibirsk, Russia (Other); I.M. Sechenov First Moscow State Medical University (Other); Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health (Other); University of Rochester (Other)
Responsible Party: Principal Investigator, Evgeny Pokushalov, Director for research and development, Center of Personalized Medicine, Pirogova
Other Study IDs: 20210308
Record Dates: First submitted 2021-03-08; First posted 2021-03-10 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Adherence to Personalized EBM Antihypertensive Drug Prescriptions for Patients With Hypertension and Comorbidities in Everyday Clinical Practice

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- By CDSS (MedicBK) Analysis
  Interventions: Drug: antihypertensive therapy
- General practice
  Interventions: Drug: antihypertensive therapy

INTERVENTIONS:
Drug: antihypertensive therapy — Personalized evidence-based antihypertensive therapy in patients with comorbidities

SUMMARY:
A retrospective analysis

DETAILED DESCRIPTION:
This retrospective study will be performed using all-Russian nationwide database of anonymized medical health claims and administrative data. The database holds information on diagnoses, patient data, medications, results of examinations, laboratory values, and genomic information, visits, follow up and outcomes. Participating health care organizations include a mix of hospital, primary care, and specialty treatment providers spanning a wide range of geographies, age groups, and income levels.

This study will analyze of outcomes according to comorbidity and antihypertensive drug prescriptions. The study will include patients who were first diagnosed with hypertension, attended the hospital as an outpatient due to hypertension, and received their antihypertensive prescription as an outpatient. To be eligible for inclusion, patients must have had comorbidities and outpatient visits or hospitalizations (for any indication) during the 3-years. The study will focused on comorbidities for choice of antihypertensive drug therapy: diabetes mellitus, dyslipidemia, gout/hyperuricemia, heart diseases, cerebrovascular diseases, and renal diseases.

We going to analyze the EMR of patients who had hypertension and comorbidities by CDSS (MedicBK) utilizing a core laboratory.

ELIGIBILITY:
Inclusion Criteria:

patients who were first diagnosed with hypertension, attended the hospital as an outpatient due to hypertension, and received their antihypertensive prescription as an outpatient. To be eligible for inclusion, patients had to have comorbidities and outpatient visits or hospitalizations (for any indication) during the 3-years.

Exclusion Criteria:

No

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with hypertension and comorbidities
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
The percentage of personalized evidence-based medicine recommendations | 3-year
  The percentage of personalized EBM recommendations acted on by clinicians for antihypertensive therapy in patients with comorbidities. All discrepancies between routine and CDSS-recommended treatment resulting in frame of guideline-based therapy and personalized EBM therapy will be adjudicated by core laboratory.

SECONDARY OUTCOMES:
3-year FU outcomes | 3-year
  Outcomes for stroke, coronary heart disease, heart failure, cardiovascular death, all cause death and the composite endpoints in relation to whether they were personalized EBM treatment or general practice.
Quantify the performance of the CDSS (MedicBK) algorithm | 3-year
  Quantify the performance of the CDSS (MedicBK) algorithm for presents treatment suggestions in frame of guideline-based therapy and personalized EBM therapy: the sensitivity, specificity, NPV, and PPV
Predictors | 3-year
  Predictors of guideline-based and personalized EBM adherence

CONTACTS AND LOCATIONS:
Overall Officials: Evgeny Pokushalov, Prof. MD PhD, Principal Investigator — Center for New Medical Technologies, Novosibirsk, Russia
Locations (1):
- Evgeny Pokushalov, Novosibirsk, Russia

IPD SHARING:
Plan to Share IPD: No